CLINICAL TRIAL: NCT00381238
Title: An Open-label Extension to Study 49653/461, to Assess the Long-term Safety of Rosiglitazone (Extended Release Tablets) in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Open-Label Extension Assessing Long-Term Safety Of Rosiglitazone In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA104617
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Rosiglitazone
MeSH Terms: conditions — Alzheimer Disease | interventions — Rosiglitazone

ARMS (1):
- rosiglitazone (Experimental): Extended Release Tablets
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — Extended Release Tablets

SUMMARY:
This is an open-label extension to study 49653/461, to assess the long-term safety of rosiglitazone (extended release tablets) in subjects with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion criteria:

* Male or female subject who has successfully completed the 12 Month Visit of 49653/461 (12 months of treatment) without tolerability issues, where in the opinion of the subject and of the investigator, it will be beneficial to continue treatment with RSG XR.
* Female subjects must be post-menopausal (i.e. >6 months without menstrual period), surgically sterile, or if of child-bearing potential, using effective contraceptive measures (oral contraceptives, Norplant, Depo-Provera, an intra-uterine device (IUD) a diaphragm with spermicide or a condom with spermicide). Women of childbearing potential must use effective contraceptive measures throughout the study and for 30 days after discontinuing study medication. The subject and their caregiver must ensure that the subject will continuously use contraceptive measures throughout the duration of the study.
* Subject is willing to participate in the extension study and has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative[1].[1] Where this is in accordance with local laws, regulations and ethics committee policy.
* Caregiver has provided full written informed consent on his or her own behalf prior to the performance of any protocol-specified procedure.

Exclusion criteria:

* Subject had a serious adverse experience (SAE) or clinically significant laboratory abnormality during 49653/461, which in the opinion of the investigator could have been attributable to study medication, and which is ongoing at the end of 49653/461.
* The subject is felt by the investigator to be unsuitable (on the basis of health, compliance, caregiver availability, or for any other reason) for inclusion in the study based on the entry criteria for the primary study, 49653/461 (exclusive of the age criteria which may not be applicable to some of the subjects).
* The subject experienced a significant cardiovascular event during 49653/461 (e.g. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia), unless a thorough cardiovascular evaluation has been performed which confirms that the subject does not have congestive heart failure, and is clinically stable.
* Treatment with a cholinesterase inhibitor, selegiline, memantine or any other treatment for cognitive symptoms/AD is initiated at the end of 49653/461.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-06-20; Primary Completion 2009-02-01 (Actual); Study Completion 2009-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (6):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Belmont, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Durham, North Carolina
- GSK Investigational Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA104617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 20 June 2006 to 03 February 2009, at seven centers in Canada and United States. This was an extension study, with a total of 33 participants with mild to moderate Alzheimer's disease, recruited in the study, who had completed 12-months of treatment in 49653/461 study.
Groups:
- RSG XR, 8 mg: The study duration was of 50-week (Wk), which comprised of a 48-Wk open-label treatment phase and a 2-Wk follow-up phase. During the treatment phase (48-Wk) the eligible participants received Rosiglitazone (RSG) extended release (XR), 4 milligram (mg) tablets once daily (od), orally in the morning for the first 4 Wks, which was followed by 8 mg od, orally in the morning for further 44 Wks of treatment.
Period: Overall Study
Arm/Group | RSG XR, 8 mg
Started | 33
Completed | 21
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy | 2
Not completed — Withdrew by physician | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Groups:
- RSG XR, 8 mg: The study duration was of 50-Wk, which comprised of a 48-Wk open-label treatment phase and a 2-Wk follow-up phase. During the treatment phase (48-Wk) the eligible participants received RSG XR, 4 mg tablets od, orally in the morning for the first 4 Wks, which was followed by 8 mg od, orally in the morning for further 44 Wks of treatment.
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 1
  White - White/Caucasian/European Heritage | 31
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE's)
Description: An AE was defined as any untoward medical occurrence or clinical investigation in a participant, temporally associated with the use of a medicinal product, whether or not, considered related to the medicinal product. For marketed medicinal products, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. The number of participants with all AEs, drug related AEs, serious adverse events (SAEs), AE leading to permanent (prm) discontinuation (disc) of study drug or withdrawal were reported.
Time Frame: From start of study medication (Wk 0) to Wk 50
Population: All subject population, is defined as all the participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participants
  All AEs | 25
  SAEs | 2
  Drug related AEs | 8
  AE leading to prm disc of study drug or withdrawal | 3

2. Secondary Outcome: Mean Change From Baseline in Mini Mental State Examination (MMSE) Total Score
Description: The MMSE, is a score scale which consists of 11 tests of orientation (to time and place), memory (recent and immediate), concentration, language and praxis. The scoring ranged from 0 to 30, with lower scores indicative of greater cognitive impairment (more severe disease) and higher scores indicative less cognitive impairment (less severe disease). The total score was calculated by summing the scores from each of the tests. The investigator questioned the participants individually with set of questions and scored the participant, based on his performance. The baseline was defined as Wk 0. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values.
Time Frame: From baseline to Wk 48
Population: Intent to treat (ITT). The ITT population consisted of all participants in the safety population who also had at least one post-dose efficacy assessment within this study.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 21
score on scale | -4.5 (4.07)

3. Secondary Outcome: Number of Participants With SAEs
Description: An SAE, is any untoward medical occurrence, that at any dose may result in death, is life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability or incapacity, is congenital anomaly or birth defect, and medically important events. The number of participants with any SAE, were reported.
Time Frame: From start of study medication (Wk 0) to Wk 50
Population: All subject population
Measure: Number; unit: participants
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participants | 2

4. Secondary Outcome: Number of Participants With AE of Peripheral Edema by Grade
Description: Participants with AE of peripheral edema were evaluated. The test was performed by firmly pressing the thumb anterior to the participants ankle until further pressure produced no greater indentation. The depth of the pit was estimated and it was graded using below 5 point scale; where estimated depth of indentation corresponded to a particular grade (G). G 0 as depth of <1 millimeter (mm); G1 as depth of 1-2 mm; G2 as depth of 3-5 mm; G3 as depth of 6-10 mm; and G4 as depth of > 10 mm. The data for only the participants who had peripheral edema on more than one visit, then their most severe G were presented.
Time Frame: Up to Wk 50
Population: All subject population
Measure: Number; unit: participants
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participants
  Participants with G0 peripheral edema | 28
  Participants with G1 peripheral edema | 3
  Participants with G2 peripheral edema | 2

5. Secondary Outcome: Mean Change From Baseline in Vital Signs- Systolic and Diastolic Blood Pressure
Description: Participants systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured in mm of mercury (mmHg). These were collected after the participant sat quietly for at least five minutes. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values.
Time Frame: Baseline (Wk 0) to Wk 50
Population: All subject population. 'n' is participants available at the particular time of assessment which were included in analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
mmHg
  DBP, Wk 2: number analyzed (Participants) | 27
  DBP, Wk 2 | -1.1 (8.31)
  SBP, Wk 2: number analyzed (Participants) | 27
  SBP, Wk 2 | 1.7 (14.56)
  DBP, Wk 4: number analyzed (Participants) | 32
  DBP, Wk 4 | -1.8 (9.25)
  SBP, Wk 4: number analyzed (Participants) | 32
  SBP, Wk 4 | -1.3 (12.91)
  DBP, Wk 8: number analyzed (Participants) | 32
  DBP, Wk 8 | 0.3 (8.19)
  SBP, Wk 8: number analyzed (Participants) | 32
  SBP, Wk 8 | 3.2 (12.96)
  DBP, Wk 16: number analyzed (Participants) | 30
  DBP, Wk 16 | -2.0 (9.69)
  SBP, Wk 16: number analyzed (Participants) | 30
  SBP, Wk 16 | -1.4 (13.94)
  DBP, Wk 24: number analyzed (Participants) | 28
  DBP, Wk 24 | -2.6 (10.22)
  SBP, Wk 24: number analyzed (Participants) | 28
  SBP, Wk 24 | 3.2 (17.96)
  DBP, Wk 32: number analyzed (Participants) | 24
  DBP, Wk 32 | -0.9 (7.96)
  SBP, Wk 32: number analyzed (Participants) | 24
  SBP, Wk 32 | 4.7 (12.59)
  DBP, Wk 40: number analyzed (Participants) | 23
  DBP, Wk 40 | -2.7 (10.10)
  SBP, Wk 40: number analyzed (Participants) | 23
  SBP, Wk 40 | 1.6 (13.96)
  DBP, Wk 48: number analyzed (Participants) | 21
  DBP, Wk 48 | -3.7 (10.13)
  SBP, Wk 48: number analyzed (Participants) | 21
  SBP, Wk 48 | 1.0 (13.72)

6. Secondary Outcome: Mean Change From Baseline in Vital Signs-heart Rate (HR)
Description: The HR for the participant's, were collected after the participant sat quietly for at least five minutes. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. The HR was measured in beats per minute (bpm).
Time Frame: Baseline (Wk 0) to Wk 50
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
bpm
  HR, Wk 2: number analyzed (Participants) | 27
  HR, Wk 2 | 1.8 (5.70)
  HR, Wk 4: number analyzed (Participants) | 32
  HR, Wk 4 | 1.2 (10.20)
  HR, Wk 8: number analyzed (Participants) | 32
  HR, Wk 8 | 1.0 (12.72)
  HR, Wk 16: number analyzed (Participants) | 30
  HR, Wk 16 | 0.3 (12.53)
  HR, Wk 24: number analyzed (Participants) | 28
  HR, Wk 24 | 1.5 (13.24)
  HR, Wk 32: number analyzed (Participants) | 24
  HR, Wk 32 | -0.2 (12.34)
  HR, Wk 40: number analyzed (Participants) | 23
  HR, Wk 40 | 1.9 (15.29)
  HR, Wk 48: number analyzed (Participants) | 21
  HR, Wk 48 | 0.1 (7.57)

7. Secondary Outcome: Number of Participants With Vital Signs of Clinical Concern.
Description: The data for number of participants with vital sign data, outside the range of potential clinical concern for SBP, DBP, HR and body weight were reported. The values as of potential clinical concern were 'both' outside of reference range or met a change from baseline criterion. The RR, for SBP was 90-140 mmHg for which the increase from baseline was reported to be >= 40 mmHg and decrease from baseline reported as >=30 mmHg; the RR for DBP was 50-90 mmHg for which the increase from baseline was reported to be >= 30 mmHg and decrease from baseline reported as >=20 mmHg; and the RR, for HR was 50-100 bpm for which the increase from baseline was reported to be >= 30 bpm and the decrease from baseline reported as >=30 bpm. The data of number of participants with > clinical concern range (CCR) or < CCR were reported.
Time Frame: Up to Wk 50
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participants
  DBP >CCR, Wk 0 | 1
  DBP <CCR, Wk 4: number analyzed (Participants) | 32
  DBP <CCR, Wk 4 | 1
  DBP >CCR, Wk 24: number analyzed (Participants) | 28
  DBP >CCR, Wk 24 | 1
  DBP <CCR, Wk 48: number analyzed (Participants) | 21
  DBP <CCR, Wk 48 | 1
  SBP >CCR, Wk 0 | 4
  SBP <CCR, Wk 0 | 1
  SBP >CCR, Wk 2: number analyzed (Participants) | 27
  SBP >CCR, Wk 2 | 5
  SBP >CCR, Wk 4: number analyzed (Participants) | 32
  SBP >CCR, Wk 4 | 4
  SBP <CCR, Wk 4: number analyzed (Participants) | 32
  SBP <CCR, Wk 4 | 1
  SBP >CCR, Wk 8: number analyzed (Participants) | 32
  SBP >CCR, Wk 8 | 5
  SBP >CCR, Wk 16: number analyzed (Participants) | 30
  SBP >CCR, Wk 16 | 1
  SBP >CCR, Wk 24: number analyzed (Participants) | 28
  SBP >CCR, Wk 24 | 3
  SBP >CCR, Wk 32: number analyzed (Participants) | 24
  SBP >CCR, Wk 32 | 5
  SBP >CCR, Wk 40: number analyzed (Participants) | 23
  SBP >CCR, Wk 40 | 7
  SBP >CCR, Wk 48: number analyzed (Participants) | 21
  SBP >CCR, Wk 48 | 1
  HR >CCR, Wk 0 | 1
  HR <CCR, Wk 4: number analyzed (Participants) | 32
  HR <CCR, Wk 4 | 1
  HR <CCR, Wk 8: number analyzed (Participants) | 32
  HR <CCR, Wk 8 | 1
  HR <CCR, Wk 16: number analyzed (Participants) | 30
  HR <CCR, Wk 16 | 1
  HR >CCR, Wk 40: number analyzed (Participants) | 23
  HR >CCR, Wk 40 | 1
  HR <CCR, Wk 40: number analyzed (Participants) | 23
  HR <CCR, Wk 40 | 1

8. Secondary Outcome: Mean Change From Baseline in Vital Signs- Weight
Description: The weight for the participant, was measured without wearing shoes and with light clothing. There was no particular RR, reported for weight; however, the increase from baseline was reported to be >=7 % and the decrease also reported as >=7 %. The values as of potential clinical concern were 'both' outside of RR, or met a change from baseline criterion.
Time Frame: Baseline (Wk 0) to Wk 50
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
kilograms
  Weight, Wk 2: number analyzed (Participants) | 27
  Weight, Wk 2 | -0.4 (1.42)
  Weight, Wk 4: number analyzed (Participants) | 32
  Weight, Wk 4 | -0.0 (1.93)
  Weight, Wk 8: number analyzed (Participants) | 32
  Weight, Wk 8 | 0.3 (2.12)
  Weight, Wk 16: number analyzed (Participants) | 30
  Weight, Wk 16 | 0.2 (3.18)
  Weight, Wk 24: number analyzed (Participants) | 28
  Weight, Wk 24 | 0.3 (3.21)
  Weight, Wk 32: number analyzed (Participants) | 24
  Weight, Wk 32 | 0.3 (3.97)
  Weight, Wk 40: number analyzed (Participants) | 23
  Weight, Wk 40 | 0.4 (3.25)
  Weight, Wk 48: number analyzed (Participants) | 21
  Weight, Wk 48 | 0.0 (2.91)

9. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Clinical Concern
Description: The data for participants for clinical parameters, with values only of potential clinical concern (PCI) were reported for creatine, creatinine kinase(CK), urea and glucose. Creatinine(unit: micromoles per litre) : low concern and high concern values were considered as 22 absolute value (AB) (<50% lower limit of RR ) and 155 (AB) (>125% upper limit of RR) respectively. CK (unit: international unit per litre ): low concern value and high concern values was none and 1.25 respectively. Glucose (unit: millimole per litre): low concern and high concern values were considered as 3.6 (AB) and 7.8 (AB) respectively.
Time Frame: Up to Wk 50
Population: All subjects population. 'n' is participants available at the particular time of assessment which were included in analysis.
Measure: Number; unit: participants
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participants
  CK, Wk 8, normal: number analyzed (Participants) | 20
  CK, Wk 8, normal | 0
  CK, Wk 8, high: number analyzed (Participants) | 20
  CK, Wk 8, high | 1
  CK, Wk 16, normal: number analyzed (Participants) | 21
  CK, Wk 16, normal | 0
  CK, Wk 16, high: number analyzed (Participants) | 21
  CK, Wk 16, high | 1
  CK, Wk 24, normal: number analyzed (Participants) | 26
  CK, Wk 24, normal | 0
  CK, Wk 24, high: number analyzed (Participants) | 26
  CK, Wk 24, high | 1
  CK, Wk 32, normal: number analyzed (Participants) | 21
  CK, Wk 32, normal | 0
  CK, Wk 32, high: number analyzed (Participants) | 21
  CK, Wk 32, high | 1
  CK, Wk 40, normal: number analyzed (Participants) | 23
  CK, Wk 40, normal | 0
  CK, Wk 40, high: number analyzed (Participants) | 23
  CK, Wk 40, high | 2
  Creatinine, Wk 8, normal: number analyzed (Participants) | 20
  Creatinine, Wk 8, normal | 0
  Creatinine, Wk 8, high: number analyzed (Participants) | 20
  Creatinine, Wk 8, high | 1
  Creatinine, Wk 8, low: number analyzed (Participants) | 20
  Creatinine, Wk 8, low | 0
  Creatinine, Wk 16, normal: number analyzed (Participants) | 21
  Creatinine, Wk 16, normal | 0
  Creatinine, Wk 16, high: number analyzed (Participants) | 21
  Creatinine, Wk 16, high | 2
  Creatinine, Wk 16, low: number analyzed (Participants) | 21
  Creatinine, Wk 16, low | 0
  Creatinine, Wk 24, normal: number analyzed (Participants) | 26
  Creatinine, Wk 24, normal | 0
  Creatinine,Wk 24, high: number analyzed (Participants) | 26
  Creatinine,Wk 24, high | 1
  Creatinine, Wk 24, low: number analyzed (Participants) | 26
  Creatinine, Wk 24, low | 0
  Creatinine, Wk 32, normal: number analyzed (Participants) | 21
  Creatinine, Wk 32, normal | 0
  Creatinine,Wk 32, high: number analyzed (Participants) | 21
  Creatinine,Wk 32, high | 1
  Creatinine, Wk 32, low: number analyzed (Participants) | 21
  Creatinine, Wk 32, low | 0
  Glucose, Wk 0, normal: number analyzed (Participants) | 19
  Glucose, Wk 0, normal | 0
  Glucose, Wk 0, high: number analyzed (Participants) | 19
  Glucose, Wk 0, high | 1
  Glucose, Wk 0, low: number analyzed (Participants) | 19
  Glucose, Wk 0, low | 0
  Urea, Wk 0, normal: number analyzed (Participants) | 11
  Urea, Wk 0, normal | 0
  Urea, Wk 0, high: number analyzed (Participants) | 11
  Urea, Wk 0, high | 1

10. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Clinical Concern-lipids
Description: Participant data for clinical concern lipid parameters for Total cholesterol, high density lipoprotein, low density lipoprotein, triglycerides was to be collected. However this data was not collected.
Time Frame: Up to Wk 50
Population: All subject population. The data for 'The number of participants with clinical chemistry parameters of clinical concern- Lipids' was not collected.
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participant's With Hematology Parameters of Clinical Concern
Description: Participant data for clinical concern hematology parameters, were reported for hematocrit (Hct) (unit:1): low concern (LC) and high concern (HC) values as 0.8 and 1.2 respectively, hemoglobin (Hb) (unit: gram per deciliter): LC and HC values as value for female (F) 10 (AB) , value for male (M) 11; and value for F 16.5 (AB), value for M 18 respectively; lymphocytes absolute(LA) (unit: giga cells per litre [GI/L]) : LC and HC value as 0.75 and 1.5 respectively; monocytes absolute (MA) (unit: GI/L) LC and HC value as 0.75 and 2 respectively, platelet count (PC) (unit: x103/mm3): LC and HC value as 100 (AB) and 500(AB) respectively, red blood cell count (RBC) (unit: x106 micro litre): LC and HC value as 0.8 and 1.2 respectively, segmented neutrophils absolute (SNA) (unit: GI/L) LC and HC value as 0.75 and 1.3 respectively, total neutrophils absolute (TNA) (unit : GI/L) LC and HC value as 0.75 and 1.5 respectively; White blood cell (WBC) (unit: GI/L) LC and HC value as 3 and 15.
Time Frame: Up to Wk 50
Population: as for outcome 9
Measure: Number; unit: participant
Arm/Group | RSG XR, 8 mg
Number analyzed (Participants) | 33
participant
  Hct, Wk 32, normal: number analyzed (Participants) | 21
  Hct, Wk 32, normal | 0
  Hct, Wk 32, high: number analyzed (Participants) | 21
  Hct, Wk 32, high | 0
  Hct, Wk 32, low: number analyzed (Participants) | 21
  Hct, Wk 32, low | 1
  Hb, Wk 8, normal: number analyzed (Participants) | 28
  Hb, Wk 8, normal | 0
  Hb, Wk 8, high: number analyzed (Participants) | 28
  Hb, Wk 8, high | 0
  Hb, Wk 8, low: number analyzed (Participants) | 28
  Hb, Wk 8, low | 1
  Hb, Wk 24, normal: number analyzed (Participants) | 28
  Hb, Wk 24, normal | 0
  Hb, Wk 24, high: number analyzed (Participants) | 28
  Hb, Wk 24, high | 0
  Hb, Wk 24, low: number analyzed (Participants) | 28
  Hb, Wk 24, low | 1
  Hb, Wk 32, normal: number analyzed (Participants) | 21
  Hb, Wk 32, normal | 0
  Hb, Wk 32, high: number analyzed (Participants) | 21
  Hb, Wk 32, high | 0
  Hb, Wk 32, low: number analyzed (Participants) | 21
  Hb, Wk 32, low | 1
  Hb, Wk 40, normal: number analyzed (Participants) | 23
  Hb, Wk 40, normal | 0
  Hb, Wk 40, high: number analyzed (Participants) | 23
  Hb, Wk 40, high | 0
  Hb, Wk 40, low: number analyzed (Participants) | 23
  Hb, Wk 40, low | 1
  Hb,Wk 48, normal: number analyzed (Participants) | 19
  Hb,Wk 48, normal | 0
  Hb, Wk 48, high: number analyzed (Participants) | 19
  Hb, Wk 48, high | 0
  Hb,Wk 48, low: number analyzed (Participants) | 19
  Hb,Wk 48, low | 1
  LA, Wk 8, normal: number analyzed (Participants) | 28
  LA, Wk 8, normal | 0
  LA, Wk 8, high: number analyzed (Participants) | 28
  LA, Wk 8, high | 0
  LA, Wk 8, low: number analyzed (Participants) | 28
  LA, Wk 8, low | 1
  LA, Wk 24, normal: number analyzed (Participants) | 28
  LA, Wk 24, normal | 0
  LA, Wk 24, high: number analyzed (Participants) | 28
  LA, Wk 24, high | 0
  LA, Wk 24, low: number analyzed (Participants) | 28
  LA, Wk 24, low | 1
  MA, Wk 0, normal,: number analyzed (Participants) | 19
  MA, Wk 0, normal, | 0
  MA, Wk 0, high: number analyzed (Participants) | 19
  MA, Wk 0, high | 0
  MA, Wk 0, low: number analyzed (Participants) | 19
  MA, Wk 0, low | 1
  MA, Wk 24, normal: number analyzed (Participants) | 28
  MA, Wk 24, normal | 0
  MA, Wk 24, high: number analyzed (Participants) | 28
  MA, Wk 24, high | 0
  MA, Wk 24, low: number analyzed (Participants) | 28
  MA, Wk 24, low | 2
  MA, Wk 40, normal: number analyzed (Participants) | 23
  MA, Wk 40, normal | 0
  MA, Wk 40, high: number analyzed (Participants) | 23
  MA, Wk 40, high | 0
  MA, Wk 40, low: number analyzed (Participants) | 23
  MA, Wk 40, low | 2
  PC, Wk 8, normal: number analyzed (Participants) | 28
  PC, Wk 8, normal | 0
  PC, Wk 8, high: number analyzed (Participants) | 28
  PC, Wk 8, high | 0
  PC, Wk 8, low: number analyzed (Participants) | 28
  PC, Wk 8, low | 2
  PC, Wk 32, normal: number analyzed (Participants) | 21
  PC, Wk 32, normal | 0
  PC, Wk 32, high: number analyzed (Participants) | 21
  PC, Wk 32, high | 0
  PC, Wk 32, low: number analyzed (Participants) | 21
  PC, Wk 32, low | 1
  PC, Wk 40, normal: number analyzed (Participants) | 23
  PC, Wk 40, normal | 0
  PC, Wk 40, high: number analyzed (Participants) | 23
  PC, Wk 40, high | 0
  PC, Wk 40, low: number analyzed (Participants) | 23
  PC, Wk 40, low | 1
  PC, Wk 48, normal: number analyzed (Participants) | 19
  PC, Wk 48, normal | 0
  PC, Wk 48, high: number analyzed (Participants) | 19
  PC, Wk 48, high | 0
  PC, Wk 48, low: number analyzed (Participants) | 19
  PC, Wk 48, low | 1
  RBC, Wk 32, normal: number analyzed (Participants) | 21
  RBC, Wk 32, normal | 0
  RBC, Wk 32, high: number analyzed (Participants) | 21
  RBC, Wk 32, high | 0
  RBC, Wk 32, low: number analyzed (Participants) | 21
  RBC, Wk 32, low | 1
  SNP, Wk 8, normal: number analyzed (Participants) | 28
  SNP, Wk 8, normal | 0
  SNP, Wk 8, high: number analyzed (Participants) | 28
  SNP, Wk 8, high | 0
  SNP, Wk 8, low: number analyzed (Participants) | 28
  SNP, Wk 8, low | 1
  SNP, Wk 24, normal: number analyzed (Participants) | 28
  SNP, Wk 24, normal | 0
  SNP, Wk 24, high: number analyzed (Participants) | 28
  SNP, Wk 24, high | 0
  SNP, Wk 24, low: number analyzed (Participants) | 28
  SNP, Wk 24, low | 1
  TNA, Wk 8, normal: number analyzed (Participants) | 28
  TNA, Wk 8, normal | 0
  TNA, Wk 8, high: number analyzed (Participants) | 28
  TNA, Wk 8, high | 0
  TNA, Wk 8, low: number analyzed (Participants) | 28
  TNA, Wk 8, low | 1
  TNA, Wk 24, normal: number analyzed (Participants) | 28
  TNA, Wk 24, normal | 0
  TNA, Wk 24, high: number analyzed (Participants) | 28
  TNA, Wk 24, high | 0
  TNA, Wk 24, low: number analyzed (Participants) | 28
  TNA, Wk 24, low | 1
  WBC, Wk 8, normal: number analyzed (Participants) | 28
  WBC, Wk 8, normal | 0
  WBC, Wk 8, high: number analyzed (Participants) | 28
  WBC, Wk 8, high | 0
  WBC, Wk 8, low: number analyzed (Participants) | 28
  WBC, Wk 8, low | 2
  WBC, Wk 16, normal: number analyzed (Participants) | 31
  WBC, Wk 16, normal | 0
  WBC, Wk 16, high: number analyzed (Participants) | 31
  WBC, Wk 16, high | 0
  WBC, Wk 16, low: number analyzed (Participants) | 31
  WBC, Wk 16, low | 2

ADVERSE EVENTS:
Time Frame: From start of study medication (Wk 0) to Wk 50
Description: All subject population was used
Arm/Group | RSG XR, 8 MG
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR, 8 MG (N=33)
Fall (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR, 8 MG (N=33)
Oedema peripheral (General disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Haematoma (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.